CLINICAL TRIAL: NCT00742703
Title: Study of the Effects of a Mineralized Water Ingestion Upon Lipidic Absorption Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Multimed (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 9808; IDRCB: 2008-A00743-52
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Moderated Cholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Mineralized water
- 2 (Active Comparator)
  Interventions: Other: Low mineralized water

INTERVENTIONS:
Other: Mineralized water
  Arms: 1
Other: Low mineralized water
  Arms: 2

SUMMARY:
The principal objective of this research is the evaluation of the effect of mineralized water consumption upon evolution of LDL Cholesterol and triglycerides, compared to a low mineralized water consumption.

ELIGIBILITY:
Inclusion Criteria:

* BMI included between 18.5 and 25 kg/m²
* non smoking
* moderated hypercholesterolemia

Exclusion Criteria:

* food allergy
* diabetes
* high blood pressure
* kidney deficiency
* thyroid deficiency
* metabolism deficiency

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-08

PRIMARY OUTCOMES:
Blood LDL Cholesterol rate. | Day-1, day-56, day-63, day-119 of study
Post-prandial blood triglycerides rate. | Day-1, day-56, day-63, day-119 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Zaïr Yassine, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Nantes, France